CLINICAL TRIAL: NCT01960920
Title: Effects of Air Pollution Exposure Reduction by Filter Mask on Heart Failure: a Prospective Randomized Double-blind Controlled Trial
Brief Title: Effects of Air Pollution Exposure Reduction by Filter Mask on Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); LABORATÓRIO DE INSUFICIÊNCIA CARDÍACA E TRANSPLANTE INCOR/HCFMUSP (Unknown); LABORATÓRIO DE POLUIÇÃO ATMOSFÉRICA EXPERIMENTAL (LPAE/ FMUSP). (Unknown)
Responsible Party: Principal Investigator, Jefferson Luis Vieira, MD, InCor Heart Institute
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 3439/10/028; 2010/50150-0 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Exposure to Pollution; Heart Failure
Keywords: Air Pollution; Heart Failure; Endothelium; Autonomic Dysfunction; Cardiopulmonary Exercise Test
MeSH Terms: conditions — Heart Failure; Primary Dysautonomias | interventions — Environment, Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (Active Comparator): Dilute diesel exhaust Filtered diesel exhaust Filtered air
  Interventions: Other: Filtered diesel exhaust; Other: Unfiltered diesel exhaust; Other: Clean air
- Heart Failure patients (Experimental): Dilute diesel exhaust Filtered diesel exhaust Filtered air
  Interventions: Other: Filtered diesel exhaust; Other: Unfiltered diesel exhaust; Other: Clean air

INTERVENTIONS:
Other: Filtered diesel exhaust — Mask-filtered exposure to diesel exhaust
  Other Names: Filter Mask 8812 (www.3m.com.br)
Other: Unfiltered diesel exhaust — Diesel Exhaust Inhalation
  Other Names: Diesel Generator Toyama TD-2500 C, www.toyama.com.br
Other: Clean air — No pollution and no filter mask

SUMMARY:
Exposure to air pollution is associated with increase in cardiovascular morbidity and mortality. Controlled human exposure studies have demonstrated impaired vascular function and heart rate variability on healthy volunteers. The aim of this study is to investigate the effects of reducting diesel exhaust inhalation on endothelial function, heart rate variability and cardiopulmonary stress testing in healthy volunteers and patients with chronic heart failure, by using a filter mask.

DETAILED DESCRIPTION:
Design and setting: Double-blind randomised crossover studies in a university teaching hospital

Patients: 30 patients with stable Heart Failure (NYHA I-III) and 15 healthy volunteers

Interventions: All 45 subjects will be exposed to dilute diesel exhaust (PM2.5 of 300 mg/m3), filtered diesel exhaust (filter mask), or filtered air

Main outcome measures: Endothelial function, heart rate variability, six-minute walking test and blood samples for inflammatory factors

ELIGIBILITY:
Inclusion Criteria:

* NYHA I-III;
* Left Ventricle Ejection Fraction < 50%;
* Clinical condition stable for more than three months prior to the randomization;

Exclusion Criteria:

* Severe arterial hypertension;
* Severe Pulmonary disease;
* Patients with pace-markers;
* Patients with constrictive pericarditis;
* Severe chronic kidney disease;
* Patients with pulmonary hypertension;
* Stroke within the last six months;
* Severe hepatic disease;
* Patients with musculoskeletal limitations to exercise;
* Patients with cardiac cachexia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | six months
  Endothelial function assessment is based on an endothelially mediated arterial response at the distal phalanx of a finger, in response to a five-minute occlusion of the brachial artery. Arterial stiffness is assessed by a finger plethysmographic probe.

SECONDARY OUTCOMES:
Heart rate variability | six months
  Heart rate variability (HRV) analysis attempts to assess cardiac autonomic regulation through quantification of sinus rhythm variability. Heart rate and beat-to-beat intervals are recorded using a frequency counter Polar Electro Oy - 800 model, interfaced to a microcomputer, and assessed using standard time domain analysis.
Inflammatory Markers | 12 months
  After each exposure, we collected blood samples for inflammatory variables-including circulating leukocytes, serum C-reactive protein, B-type natriuretic peptide, Troponin and Catecholamines.
Six-minute walking test | Six months
  Exercise testing is performed on a treadmill using a modified Naughton protocol and the 6 minute walk test. Ventilation, oxygen uptake, and carbon dioxide production are monitored continuously using a respiratory mass spectrometer.

CONTACTS AND LOCATIONS:
Overall Officials: Edimar A Bocchi, pHD, Study Chair — Heart Failure Lab. Coordinator
Locations (1):
- Heart Failure Lab. Incor HCFMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Vieira JL, Guimaraes GV, de Andre PA, Cruz FD, Saldiva PH, Bocchi EA. Respiratory Filter Reduces the Cardiovascular Effects Associated With Diesel Exhaust Exposure: A Randomized, Prospective, Double-Blind, Controlled Study of Heart Failure: The FILTER-HF Trial. JACC Heart Fail. 2016 Jan;4(1):55-64. doi: 10.1016/j.jchf.2015.07.018. PMID 26738952